CLINICAL TRIAL: NCT06175949
Title: A Randomized, Double-Blind, Dose-Escalation, Placebo-Controlled Phase I Clinical Trial Assessing the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HRS-7085 Tablets Following Single and Multiple Oral Administrations, With Evaluation of Food Effects in Healthy Subjects
Brief Title: A Randomized, Double-Blind, Dose-Escalation, Placebo-Controlled Phase I Clinical Trial Investigating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Oral Doses of HRS-7085 Tablets in Healthy Subjects, With Assessment of Food Effects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7085-101
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-7085 (Experimental)
  Interventions: Drug: HRS-7085 Tablets
- HRS-7085 simulant (Placebo Comparator)
  Interventions: Drug: HRS-7085 simulant

INTERVENTIONS:
Drug: HRS-7085 Tablets — HRS-7085 Tablets, PO, 2mg、5mg、8mg、10mg、12mg、15mg, QD,
  Arms: HRS-7085
Drug: HRS-7085 simulant — PO, 2mg、5mg、8mg、10mg、12mg、15mg, QD
  Arms: HRS-7085 simulant

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-parallel-controlled, Phase I clinical trial investigating the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple oral doses of HRS-7085 tablets in healthy subjects, with assessment of food effects

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 55 years (inclusive), of any gender (each dose group should include at least two subjects of a single gender, except for the 2 mg dose group in Part 1A).
2. Body Mass Index (BMI = weight/height^2) during screening: 19 ≤ BMI < 28 kg/m^2; male weight ≥ 50.0 kg and < 90.0 kg, female weight ≥ 45.0 kg and < 90.0 kg.
3. Healthy subjects with physical examination, vital signs, and laboratory test results (including complete blood count, urinalysis, blood biochemistry, coagulation function, thyroid function), chest X-ray, 12-lead electrocardiogram, abdominal ultrasound, judged by the investigator as normal or clinically insignificant abnormalities during screening.
4. Female subjects of reproductive potential and male subjects with female partners of reproductive potential must have no plans for reproduction, sperm/egg donation for at least 3 months after the last dose and voluntarily agree to use effective contraception. Serum pregnancy test for female subjects must be negative and not in lactation.
5. Obtain informed consent before any trial-related activities begin, fully understand the purpose and significance of this trial, and be willing to comply with the trial protocol.

Exclusion Criteria:

1. Within the past year prior to screening or dosing, individuals with systemic diseases such as cardiovascular, hepatic, renal, gastrointestinal, psychiatric, neurological, or hematologic conditions, deemed by the investigator to pose potential safety risks.
2. Within the past 6 months prior to screening or dosing, individuals with a history of severe infections (such as bloodstream infections, central nervous system infections, abdominal infections, etc.), severe trauma, or major surgeries (excluding appendectomy); those planning to undergo surgery during the trial.
3. Within the past month prior to screening or dosing, individuals with a history of infections (viral, bacterial, fungal, parasitic) requiring systemic antimicrobial therapy.
4. Individuals experiencing frequent headaches, nausea, and/or vomiting with a frequency of ≥3 times per month.
5. Individuals with allergic tendencies, such as a history of asthma, atopic dermatitis, chronic urticaria, allergic rhinitis, or any known allergies to drugs or foods.
6. Within the past month prior to screening or dosing, individuals who donated blood or experienced blood loss ≥200 mL, or within the past 3 months prior to dosing, individuals who donated blood or experienced blood loss ≥400 mL.
7. As determined by the study physician, individuals with any physiological or psychological condition that may increase trial risks, affect subject compliance with the protocol, or interfere with subject completion of the trial.
8. Individuals with a smoking history within the past 3 months prior to screening (average daily smoking >5 cigarettes) or those unable to abstain from any tobacco products during the trial.
9. Within the past month prior to screening, individuals with an average daily alcohol intake exceeding 7 g for females (equivalent to approximately 200 mL of beer, 70 mL of wine, or 22 mL of spirits) or exceeding 14 g for males (equivalent to approximately 400 mL of beer, 140 mL of wine, or 45 mL of spirits); or individuals with a positive alcohol test at screening or those unable to abstain from alcohol during the trial.
10. Individuals who consumed any grapefruit-containing foods or beverages within 7 days prior to taking the study drug, or those who consumed caffeine-containing foods or beverages within 2 days prior to taking the study drug.
11. Individuals with special dietary requirements who cannot adhere to a standardized diet.
12. Individuals with a history of drug abuse or substance misuse, or those with a positive urine drug screen at screening.
13. Individuals with positive results in infectious disease screening tests (HBsAg, anti-HCV Ab, anti-TP Ab, anti-HIV Ab) at screening.
14. Individuals with alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin (TBIL) levels ≥1.5 times the upper limit of normal (ULN) at screening.
15. Within 2 weeks prior to screening or dosing, individuals who used any prescription medications, over-the-counter medications, or herbal supplements; or individuals within 5 half-lives of a drug (whichever is longer) at screening or planning to use non-study investigational drug during the trial.
16. Within the past 3 months prior to screening, individuals who participated in any other clinical trial (excluding those who failed screening) or those still within 5 half-lives of a drug (whichever is longer) at screening.
17. Within the past 3 months prior to screening, individuals who received a live vaccine or attenuated live vaccine, or those planning to receive any vaccines during the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 7 days or 20 days,

IPD SHARING:
Plan to Share IPD: Undecided